CLINICAL TRIAL: NCT07073586
Title: Protocol: Effect of Lymphovenous Anastomosis in the Treatment of Lower Limb Lymphedema - Pragmatic Assessor-Blinded Open-Label Randomized Controlled Trial (PrCT)
Brief Title: Effect of Lymphovenous Anastomosis on Lower Limb Lymphedema: Pragmatic Randomized Controlled Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Herlev and Gentofte Hospital (Other)
Responsible Party: Principal Investigator, Amar Bucan, Medical doctor, Herlev and Gentofte Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H-25012096
Record Dates: First submitted 2025-07-09; First posted 2025-07-18 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Lymphedema; Lymphoedema; Lymphoedema of Leg; Lymphedema of Leg
Keywords: Lymphovenous Anastomosis; LVA; Lower Limb Lymphedema; Leg Lymphedema; Randomized Controlled Trial; CDT; Compression Therapy
MeSH Terms: conditions — Lymphedema

STUDY DESIGN:
Intervention Model Description: Two-arm, assessor-blinded, open-label, pragmatic randomized controlled trial comparing LVA plus conservative therapy with conservative therapy alone.
Who Masked: Outcomes Assessor
Masking Description: Outcome assessors remain unaware of group allocation; participants wear adhesive bandage over potential incision sites at follow-up visits.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lymphovenous anastomosis (LVA) + Compression Therapy (Experimental): LVA + conservative care. Patient must have undergone Complete Decongestive Therapy (CDT) and comply with the compression treatment. Follow-up at 6, 12 and 24 months includes blinded assessment of L-Dex, tape and perometry volumes, DXA, lymphoscintigraphy, erysipelas incidence and LYMQOL/EQ-5D-5L scores; patency is checked by ICG-lymphography at 12 months. A subset of 10 patients with unilateral lymphedema also provides paired skin biopsies (both legs) at surgery and again 6 months postoperatively for biomarker and histological analysis.
  Interventions: Procedure: Lymphovenous Anastomosis; Other: Complete Decongestive Therapy
- Compression Therapy Alone (Active Comparator): Conservative care alone. Participants complete standard Complete Decongestive Therapy, comprising bandaging, skin care and exercise, followed by compression garments. Outcomes are assessed by the same blinded schedule as the LVA arm at baseline, 6, 12 and 24 months. Participants may elect LVA crossover after the 12-month evaluation if desired.
  Interventions: Other: Complete Decongestive Therapy

INTERVENTIONS:
Procedure: Lymphovenous Anastomosis — Microsurgical creation of multiple lymphatic-venous connections in the most affected limb under general anaesthesia.
  Arms: Lymphovenous anastomosis (LVA) + Compression Therapy
Other: Complete Decongestive Therapy — Complete Decongestive Therapy, comprising bandaging, skin care and exercise, followed by compression garments.
  Other Names: CDT

SUMMARY:
This multicentre pragmatic randomised controlled trial evaluates lymphovenous anastomosis (LVA) for lower-limb lymphedema (LLL) in Denmark. Adults with unilateral or bilateral International Society of Lymphology (ISL) stage 1-2a LLL who have completed protocol-defined Complete Decongestive Therapy (CDT) are randomised 1:1 to

Intervention arm - LVA surgery plus ongoing compression care

Control arm - Compression care only

Recruitment takes place at the Departments of Plastic Surgery, Herlev-Gentofte Hospital and Odense University Hospital. Outcomes are assessed by independent blinded staff at baseline, 6, 12 and 24 months. A biopsy substudy in ten LVA patients explores inflammatory and fibrotic changes. Primary endpoint is change in L-Dex ratio at 12 months. Secondary endpoints include limb volume, infection rate, lymphoscintigraphy findings, patient-reported outcomes, compression-garment use and anastomosis patency.

The trial follows Good Clinical Practice and General Data Protection Regulation (GDPR). Patients are covered by the Danish public patient-compensation scheme. Results will be published regardless of outcome, and control participants may opt for LVA after the 12-month visit.

DETAILED DESCRIPTION:
Lower-limb lymphedema (LLL) causes chronic swelling, pain, recurrent infections and impaired quality of life. Complete Decongestive Therapy (CDT) is standard care, yet many patients have persistent disease. Lymphovenous anastomosis (LVA) is a super-microsurgical procedure that diverts lymph into the venous system, but robust randomised evidence in LLL is lacking

This multicentre pragmatic randomised trial will test whether lymphovenous anastomosis (LVA) can reduce lower-limb lymphedema and improve life quality in adults who have completed Complete Decongestive Therapy (CDT). The study is carried out at two Danish university hospitals that routinely manage complex lymphedema. A computer system assigns participants in a 1:1 ratio to either LVA plus compression care or compression care alone. Surgeons create as many anastomoses as possible under general anaesthesia, using indocyanine green mapping to find suitable lymphatic vessels.

Adults aged 18 years or older with International Society of Lymphology stage (ISL) 1 or 2a lymphedema of one or both legs can join if they have finished CDT. Key exclusions are stage 2b or 3 disease, body-mass index (BMI) above 28, active cancer, severe medical illness, or prior lymphedema surgery.

The primary outcome is the change in L-Dex ratio, from baseline to 12 months. Secondary outcomes measured at baseline, 6, 12 and 24 months include limb volume by tape, perometry and dual-energy X-ray absorptiometry, infection frequency, lymphoscintigraphy findings, quality-of-life scores (Lymphedema Quality of Life Questionnaire (LYMQOL) and EuroQol Five Dimension Five Level (EQ-5D-5L)) and use of compression garments. At 12 months the patency of the anastomoses is checked with indocyanine green lymphography in the surgical arm. A small substudy in ten surgical participants will compare inflammatory markers and tissue structure in paired skin biopsies collected during surgery and again 6 months later.

Participants attend the clinic for baseline, 6-month and 12-month visits and return at 24 months for long-term follow-up. Conservative measures such as compression garments may continue (but not reduced in 12 months for LVA-group), but no other surgical or medical lymphedema procedures are allowed during the study period.

All data are entered into a secure electronic database and analysed according to Good Clinical Practice, the Danish Code of Conduct for Research Integrity and General Data Protection Regulation (GDPR). The regional research ethics committee has approved the protocol, and participants are covered by the Danish public patient-compensation scheme. Results will be published in peer reviewed journals no matter whether LVA shows benefit, harm or no difference.

ELIGIBILITY:
Inclusion Criteria:

* LLL International Society of Lymphology (ISL) stage 1-2a (both primary and secondary lymphedema and both unilateral and bilateral)
* Cancer-free with no recurrence for at least one year
* Age 18 or above
* Circumference of the affected leg is at least 1 cm larger than the non-lymphedema leg at the most affected site of lymphedema.
* Proficiency in Danish language, and ability to provide informed consent.
* Dermal Backflow Stage 0-4

Exclusion Criteria:

* LLL International Society of Lymphology (ISL) stage 2b-3
* Medical conditions contraindicating surgical intervention or anesthesia, such as severe heart or lung disease
* Allergy to ICG
* Ongoing infections or skin diseases in the affected limb
* Previous surgery or other treatment modalities that could interfere with the study results (previous LVA, liposuction or similar).
* Dermal Backflow Stage 5
* Active cancer
* Heart or kidney conditions that can cause leg swelling
* A BMI above 28 kg/m²
* Current smoker
* Any foreign objects in the lower extremities (e.g., metal implants, prostheses)
* Venous insufficiency Unilateral weakness in the lower extremity (e.g., after a stroke)
* Known iodine allergy (contraindication for ICG injection)
* Leg length discrepancy (anisomelia) > 1.5 cm

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2025-05-09 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2029-08 (Estimated)

PRIMARY OUTCOMES:
Change in L-Dex ratio (bioimpedance spectroscopy) at 12 months. | Baseline to 12 months
  Difference in L-Dex ratio of the most affected leg, measured with the SOZO bioimpedance device (ImpediMed). Measurements are performed by blinded assessors after 48 h without compression garments.

SECONDARY OUTCOMES:
Change in Limb Volume by Tape Measurement | Baseline, 6 months, 12 months, 24 months
  Difference in limb volume using tape measurements and calculating using formulas.
Change in Limb Volume by Perometry | Baseline, 6 months, 12 months, 24 months
  Difference in limb volume obtained with optoelectronic perometry (automatic three-dimensional scan of the leg).
Change in Limb Mass by DXA | Baseline, 6 months, 12 months, 24 months
  Difference in limb mass of the affected leg measured with dual-energy X-ray absorptiometry.
Change in Compression Garment Use | Baseline to 24 months
  Change of compression class, change in daily use, or continue/discontinue compression garments. Data collected by questionnaire.
Incidence of Erysipelas Infections | Baseline, 6 months, 12 months, 24 months
  Number of erysipelas episodes in the affected limb
Change in Lymphoedema Quality of Life Questionnaire (LYMQOL) | Baseline, 6 months, 12 months, 24 months
  Difference in total score of the Lymphoedema Quality of Life Questionnaire for lower limb lymphedema.
  Item and domain scores run from 1 to 4. Higher scores mean a worse quality of life.
  The separate "overall quality of life" item uses a 0 to 10 scale. Higher scores mean a better quality of life.
Change in EuroQol Five Dimension Five Level (EQ-5D-5L) utility index | Baseline, 6 months, 12 months, 24 months
  Using the Danish value set, scores range from -0.757 (worst imaginable health) to 1.000 (full health). Higher scores mean a better health-related quality of life
Change in Lymphoscintigraphy | Baseline, 6 mo, 12 mo, 24 mo
  Change in lymphoscintigraphy transport. Scans read by blinded nuclear-medicine specialists.

OTHER OUTCOMES:
Patency of Lymphovenous Anastomoses | 12 months
  Proportion of anastomoses that remain patent on indocyanine green (ICG) lymphography performed in the LVA group. Patency defined as visible dye passage through the anastomosis.
Change in Biomarkers in Skin Biopsies | Baseline (intra-operative) to 6 months
  Change in expression of cytokines and growth factors in paired biopsies from affected and contralateral legs of 10 LVA participants.
Change in Histological Features in Skin Biopsies | Baseline (intra-operative) to 6 months
  Difference in histology and immunohistochemistry on the same paired biopsies in paired biopsies from affected and contralateral legs of 10 LVA participants.

CONTACTS AND LOCATIONS:
Overall Officials: Lisbet Rosenkrantz Hölmich, MD, Professor, DMSc, Study Chair — Department of Plastic Surgery, Herlev and Gentofte Hospital, Denmark
Locations (2):
- Denmark (2):
  - Department of Plastic Surgery, Odense University Hospital, Odense, Fyn
  - Department of Plastic Surgery, Herlev and Gentofte Hospital, Herlev, Region Sjælland

IPD SHARING:
Plan to Share IPD: No